CLINICAL TRIAL: NCT01091376
Title: A Phase II Study of Erlotinib Combined With Radiotherapy in Patients With Non-resectable Locally Advanced Non-small Cell Lung Cancer
Brief Title: Erlotinib Combined With Radiotherapy in Patients With Non-resectable Locally Advanced Non-small Cell Lung Cancer (LA-NSCLC)
Acronym: RT0901
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Shenglin Ma, Lvhua Wang, Zhejiang Cancer Hospital; Chinese Academy of Medical Sciences Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH02
Record Dates: First submitted 2010-01-14; First posted 2010-03-24 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; EGFR-TKI; Erlotinib; Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Concomitant Erlotinib and radiotherapy (Experimental): Patients received Erlotinib and radiation therapy.
  Interventions: Drug: Erlotinib; Radiation: Thoracic radiotherapy

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150mg/day
Radiation: Thoracic radiotherapy — 60-70Gy/30-35f

SUMMARY:
Concomitant chemoradiotherapy is the standard treatment of locally advanced,non-resectable, non-small cell lung cancer (NSCLC). However,the optimal chemotherapy regimen is still controversial.The objective of this study was to evaluate the efficacy and toxicity of a concomitant treatment using Erlotinib and radiotherapy followed by Erlotinib consolidation treatment.

DETAILED DESCRIPTION:
Patients with non-resectable Non-small Cell Lung Cancer will receive thoracic radiation therapy 60-70 Gy over 30-35 fractions and concurrent with Erlotinib 150mg/day. Followed by Erlotinib 150 mg/day consolidation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven non-small cell lung cancer (squamous cell carcinoma, adenocarcinoma, large cell carcinoma and etc)
* Tumor EGFR mutation
* Presence of measurable disease by RECIST
* stage IIIA or IIIB, non-resectable
* ECOG performance status 0-2
* No prior chemotherapy, radiation therapy to chest, immunotherapy, or biologic therapy
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital.

Exclusion Criteria:

* Carcinoid tumor, small cell carcinoma of lung
* Patients with any distant metastasis
* History of another malignancy except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* Any other morbidity or situation with contraindication for radiotherapy (e.g. active infection, myocardial infarction preceding 6 months, symptomatic heart disease including unstable angina, congestive heart failure or uncontrolled arrhythmias, immunosuppressive treatment)
* Pregnant or lactating women, women who has not taken test of pregnancy (within 7 days before the first administration) and pregnant women
* Women and men of childbearing potential who have no willing of employing adequate contraception
* Tumor EGFR wild

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate (Response was analyzed according to the RECIST system, based on CT scans.) | After the thoracic radiotherapy and concurrent Erlotinib treatment
The safety (The safety was evaluated according to the National Cancer Institute Common Toxicity Criteria version 3.0.) | Every one month

SECONDARY OUTCOMES:
Progression free survival | The time from the start of treatment to diease progression
The overall survival | The time from the start of treatment to death
Quality of Life (QoL was evaluated according to the FACT-L.) | Every one month

CONTACTS AND LOCATIONS:
Overall Officials: Shenglin Ma, MD, Principal Investigator — Zhejiang Cancer Hospital; Lvhua Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China